CLINICAL TRIAL: NCT03524391
Title: Effect of Yoga Counselling on Quality of Life and Psychological Outcomes of Prostate Cancer Patients: Randomized Control Trial
Brief Title: Effect of Yoga Counselling on Quality of Life and Psychological Outcomes of Prostate Cancer Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NMP Medical Research Institute (Other)
Collaborators: Warwick Research Services (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: NMP/10123
Record Dates: First submitted 2018-05-02; First posted 2018-05-14 (Actual); Last update posted 2018-05-14 (Actual); Status verified 2018-05

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Drug Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Yoga Counselling Group (Experimental): Yoga based psychological counselling delivered individually and in group along with conventional care
  Interventions: Behavioral: Counselling based on yoga; Drug: Chemotherapy
- Usual Care Group (Active Comparator): Usual care provided to patients
  Interventions: Drug: Chemotherapy

INTERVENTIONS:
Behavioral: Counselling based on yoga — Counseling sessions were given as one-on-one and group to patients based on yoga philosophy and therapy.
  Arms: Yoga Counselling Group
Drug: Chemotherapy — Usual Care group had standard chemotherapy regimens

SUMMARY:
Cancer is second leading cause of death worldwide. The psychological issues are related to all stages of the disease affecting outcome of treatment and overall quality of life. The study evaluated the effectiveness of yoga counselling among prostate cancer patients on their quality of life and psychological outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Primary diagnosis of Prostate Cancer
* Sign a consent form allowing related information to be included in this research.

Exclusion Criteria:

* Have pre-existing diagnosed psychiatric conditions
* Currently taking psychotropic medications
* Have been diagnosed with cancer other than prostate cancer
* Evidence of active substance abuse.

Ages: 40 Years to 60 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 92 (Actual)
Dates: Start 2016-02-12 (Actual); Primary Completion 2017-01-05 (Actual); Study Completion 2017-02-25 (Actual)

PRIMARY OUTCOMES:
Anxiety and Depression | Change from baseline to 12 weeks
  Depression and anxiety as assessed by Hospital Anxiety Depression Scale

SECONDARY OUTCOMES:
Quality of Life | Change from baseline to 12 weeks
  Quality of life as assessed by WHO quality of life-BREF

CONTACTS AND LOCATIONS:
Overall Officials: Neha Sharma, PhD, Study Director — Warwick Research Services; Dhruv Singh, Principal Investigator — NMP Medical Research Institute, India

IPD SHARING:
Plan to Share IPD: Undecided